CLINICAL TRIAL: NCT00948987
Title: Mechanism Based Resistance to Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Bayer (Industry)
Responsible Party: Garret A. FitzGerald, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 801907; 0926
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Aspirin Resistance; Pharmacological Aspirin Non-responsiveness
Keywords: aspirin resistance; cardiovascular risk; prostaglandins; platelet inhibition
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspirin (Experimental): single dose of aspirin 325 mg p.o.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 325 mg enteric coated single dose p.o.

SUMMARY:
The purpose of this research is to study why some people do not respond to the benefits of aspirin therapy. The benefit of aspirin is cardioprotection, or decreasing the risk of heart attack and/or stroke. Aspirin works by disabling the platelets, part of the blood cells used in clotting, from sticking together and forming blood clots, thus protecting the heart. It has been observed that failure to respond to aspirin therapy occurs in about 10% of the general population and that despite taking aspirin everyday, this group of non- responders is not getting protection for their heart. The investigators would like to determine why and how this happens.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 55
* Subjects must be in good health as based on medical history, physical examination, vital signs, and laboratory tests.
* All subjects must be non- smoking volunteers
* Female subjects of child bearing potential must be using a medically acceptable method of contraception (oral contraception, depo-provera injection, IUD, condom with spermicide, diaphragm, cervical cap, progestin implant, abstinence, tubal ligation, oophorectomy, TAH) throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and just prior to the start of each treatment phase of the study, which must be negative at all time points.
* Subjects must be within 30% of their ideal body weight.

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects with any coagulation, bleeding or blood disorders.
* Subjects who are sensitive or allergic to aspirin as well as any of their components.
* Subjects with documented history of any gastrointestinal disorders, including bleeding ulcers.
* Subjects with any evidence of cancer.
* Subjects with a history of heart disease, including myocardial infarction, angina, coronary artery disease, any evidence of coronary artery stenosis, arrhythmias, heart failure, having had a CABG
* Subjects with renal, hepatic, respiratory, endocrine, metabolic, hematopoietic or neurological disorder.
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Subjects who have had a history of drug or alcohol abuse within the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2004-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Arachidonic acid induced platelet aggregation | 8 hours postdose

SECONDARY OUTCOMES:
Serum thromboxane B2 concentration Urinary 11-dehydro thromboxane B2 concentration Urinary 2,3 dinor-6 keto PGF1α concentration | 8 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics; Susanne Fries, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics; Tilo Grosser, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics

REFERENCES:
- [Derived] Grosser T, Fries S, Lawson JA, Kapoor SC, Grant GR, FitzGerald GA. Drug resistance and pseudoresistance: an unintended consequence of enteric coating aspirin. Circulation. 2013 Jan 22;127(3):377-85. doi: 10.1161/CIRCULATIONAHA.112.117283. Epub 2012 Dec 4. PMID 23212718